CLINICAL TRIAL: NCT00585156
Title: The Effects of Celecoxib on Bone Ingrowth in Porous Coated Titanium Ceramic Implants in Humans
Brief Title: The Effects of Celecoxib on Bone Ingrowth
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: New clinical finding with Celebrex and cardiac concerns.
Sponsor: University of Utah (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: IIR#2005-0300; IIR#2005-0300
Record Dates: First submitted 2007-12-26; First posted 2008-01-03 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Bone Ingrowth; Pain
Keywords: Celebrex, Bone Ingrowth, Pain relief
MeSH Terms: conditions — Pain | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm #1 (Experimental): Celebrex treatment group
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Celecoxib — Twelve hours prior to their first total knee surgery, patients will need to take an oral dose of Celebrex, 1 pill of 200mg. Following the patient's first total knee surgery, they will continue taking oral doses of Celebrex, 1 pill of 200 mg every twenty-four hours (200mg/day) for a two-week period.
  Other Names: Celebrex

SUMMARY:
The purpose of this study is to evaluate the effect of Celebrex on bone growth into porous coated implants, following postoperative total knee arthroplasty administration of Celebrex for pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Male VA bilateral TKA patients 18 years or older with primary OA diagnosis

Exclusion Criteria:

* Patients with osteoporosis, hypersensitivity to Celebrex, allergy to tetracycline, Sulfonamides, patient with asthma, urticaria, or allergic-type reactions to aspirin or NSAIDs.
* Patients who have had CABG.
* Patients with a history of peptic ulcer disease, duodenal ulcers.
* Female patients and patients diagnosed with unstable hypertension or hypotensive, with serum creative levels above 1.8-2.0 or diagnosed with severe renal disease.

Ages: 18 Years to 95 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Bone Ingrowth | 12 weeks

SECONDARY OUTCOMES:
Pain Score | 10 days postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Roy Bloebaum, Ph.D., Principal Investigator — Research Professor, Orthopedic Surgery
Locations (1):
- Veteran Affairs (VA) Medical Center, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Hofmann AA, Bloebaum RD, Rubman MH, Bachus KN, Plaster RL. Microscopic analysis of autograft bone applied at the interface of porous-coated devices in human cancellous bone. Int Orthop. 1992;16(4):349-58. doi: 10.1007/BF00189618. PMID 1473888
- [Background] Hofmann AA, Bloebaum RD, Koller KE, Lahav A. Does celecoxib have an adverse effect on bone remodeling and ingrowth in humans? Clin Orthop Relat Res. 2006 Nov;452:200-4. doi: 10.1097/01.blo.0000238838.18799.61. PMID 17016230